CLINICAL TRIAL: NCT03587415
Title: Serum Preptin and Amylin Levels With Respect to Body Mass Index in Polycystic Ovary
Brief Title: Serum Preptin and Amylin Levels in Polycystic Ovary Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Senol Senturk, Serum Preptin and Amylin Levels in Polycystic Ovary Syndrome Patients, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 107
Record Dates: First submitted 2018-06-12; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: amylin; obesity; polycystic ovarian syndrome; preptin
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polycyctic ovary sendrome (PCOS): these women who have PCOS, we will use their blood samples
  Interventions: Diagnostic Test: preptin and amylin level
- Healty groups: These women who have reguler menstrual cycle, no akne or hirsutism, we will use their boold samples
  Interventions: Diagnostic Test: preptin and amylin level

INTERVENTIONS:
Diagnostic Test: preptin and amylin level — we will take both of group blood samples to compare them serum preptin and amylin

SUMMARY:
Preptin and amylin are pancreatic hormones which participate in glucose homeostasis. This study aims to evaluate how serum preptin and amylin levels are altered in polycystic ovary syndrome (PCOS) patients and healthy women based on BMI groups .

DETAILED DESCRIPTION:
Materials and Methods: This is a cross-sectional review of 40 PCOS patients and 40 healthy women who were matched with respect to BMI (<25 kg/m2 and ≥25 kg/m2).

ELIGIBILITY:
Inclusion Criteria:

the patients with PCOS

Exclusion Criteria:

Cushing's syndrome 21-hydroxylase deficiency Congenital adrenal hyperplasia Thyroid dysfunction Hyperprolactinemia Diabetes Chronic cardiovascular Hepatic, renal, and hematologic diseases Malignancies Using oral contraceptives, anti-androgens, glucocorticoids, anti-hypertensives, anti-diabetics, calcium supplements and anti-obesity drugs and those who smoke or consume alcohol

-

Ages: 17 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polycystic ovary syndrome
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Serum Preptin and Amylin Levels with Respect to Body Mass Index in Polycystic Ovary Syndrome Patients | six months
  Serum Preptin and Amylin Levels will compare between groups

CONTACTS AND LOCATIONS:
Overall Officials: Senol sentürk, PhD, Study Director — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)